CLINICAL TRIAL: NCT00686387
Title: Establishment of a Brain and Spinal Tumor Tissue Bank and Clinical Data Repository for Identifying Molecular Markers of Clinical Outcome
Brief Title: Establishment of a Brain and Spinal Tumor Tissue Bank
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Kuo-Sheng Hung, MD,, Taipei Medical University-Wan Fang Hospital
Other Study IDs: 2008WFCRC-01
Record Dates: First submitted 2008-05-26; First posted 2008-05-29 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Glioblastoma Multiforme; Glioma; Neuroectodermal Tumors
Keywords: Tissue Bank; Glioblastoma Multiforme; NAT2; EGFR; MGMT; Brain and Spinal TumorGliomas
MeSH Terms: conditions — Glioblastoma; Glioma; Neuroectodermal Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, Fresh tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to establish a Brain and Spinal Tumor Tissue/Specimen repository to serve as a resource for current and future scientific studies.

DETAILED DESCRIPTION:
Glioblastoma multiforme (GBM) is the most common and lethal primary Brain and Spinal Tumor in adults. It is nearly uniformly fatal, with a median survival of approximately one year, despite modern treatment modalities. Efforts to understand why some patients live longer or shorter than the average may provide insights into the biology of these neoplasms. For years, researchers have tried to identify independent predictors that could help in treatment planning. With the recent interest in molecular biology and molecular genetics, tumor markers are now being examined as potential predictors. A marker that could predict tumor response to therapy, the likelihood of recurrence, and survival would thus be quite useful.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a suspected or confirmed diagnosis of Brain and Spinal Tumor
* Age greater than 20
* Signed consent

Exclusion Criteria:

* Known HIV infection
* Any other clinical condition which, in the opinion of the principal investigator, would not allow completion of this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurosurgery clinic or oncology clinic in Wan Fang Hospital
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2008-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Collect, annotate, and store fresh frozen specimens of normal tissue, tumors, and pre-malignant lesions for biological investigation. | 5 years

SECONDARY OUTCOMES:
Collect, process, and store serum, plasma and isolate lymphocytes from blood drawn from patients with Brain and Spinal Tumor | 5 years
Establish a database to link materials acquisition, pathologic, and clinical information on patients who participate in the protocol | 5 years
To utilize the clinical database to perform clinical and pathological correlation with the results of current and future scientific studies | 5 years
To evaluate various NAT2, EGFR and MGMT for evidence of genomic and biochemical activation | 5 years
To test the effect of small molecule inhibitors on the activation of wild-type and mutant NAT2, EGFR, MGMT and/or other potential molecular targets | 5 years
To correlate tumor genotype and signaling abnormalities with clinical response to NAT2, EGFR, MGMT and/or other potential molecular targets inhibitors | 5 years
Analysis of laboratory findings in relationship to patient demographics and clinical course | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Sheng Hung, MD, PhD, Principal Investigator — Taipei Medical University-Wan Fang Hospital
Locations (1):
- Taipei Medical University-Wan Fang Hospital, Taipei, Taiwan